CLINICAL TRIAL: NCT04505995
Title: Efficacy of Concomitant Use of Azacitidine and Homoharringtonine in Children With Juvenile Myelomonocytic Leukemia
Brief Title: Azacitidine and Homoharringtonine in JMML
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Air Force Military Medical University, China (Other)
Collaborators: Qilu Hospital of Shandong University (Other); Taian City Central Hospital (Other); The Affiliated Hospital of Qingdao University (Other); The Second Hospital of Hebei Medical University (Other); Children's Hospital of Hebei Province (Other)
Responsible Party: Principal Investigator, Lipeng Liu, Dr, Air Force Military Medical University, China
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: JMML-CAMS-2020
Record Dates: First submitted 2020-08-06; First posted 2020-08-10 (Actual); Last update posted 2020-08-10 (Actual); Status verified 2020-08

CONDITIONS: JMML
MeSH Terms: interventions — Azacitidine; Homoharringtonine

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Intervention group (Experimental)
  Interventions: Drug: Azacitidine and homoharringtonine

INTERVENTIONS:
Drug: Azacitidine and homoharringtonine — Concommitant use of azacitidine and homoharringtonine

SUMMARY:
Juvenile myelomonocytic leukemia (JMML) has a poor prognosis in general, with hematopoietic stem cell transplant (HSCT) remaining the standard of care for cure. Azacitidine and homoharringtonine, which exhibited a anticancer mechanism and has been widely used in patients with relapse/refractory acute myeloid leukemia (AML). However, the efficacy of these agents has not been elucidated in children with JMML. The primary objective is to assess the treatment effect on response rate in this subject population.

ELIGIBILITY:
Inclusion Criteria:

* Newly diagnosed JMML, with PB and BM confirming diagnosis prior to informed consent signature, with one of the following:

  1. somatic mutation in PTPN11
  2. somatic mutation in KRAS
  3. somatic mutation in NRAS and HbF % > 5x normal value for age
  4. clinical diagnosis of neurofibromatosis Type 1.

Exclusion Criteria:

* 1. Any condition that would prevent the subject from participating in the study.

  2. Any condition including the presence of laboratory abnormalities, which places the subject at unacceptable risk if participated in the study.

  3. Any condition that confounds the ability to interpret data from the study.

Ages: 1 Month to 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 30 (Estimated)
Dates: Start 2020-01-01 (Actual); Primary Completion 2023-01-01 (Estimated); Study Completion 2025-01-01 (Estimated)

PRIMARY OUTCOMES:
Juvenile Myelomonocytic Leukemia (JMML) response rate at end of 4 Months | Up to 4 Months
  Defined as proportion of patients with sustained clinical complete remission [cCR] or clinical partial remission [cPR] according to the International JMML response criteria in Niemeyer 2014 at 3 months (28 days cycles). Response must be sustained for at least 4 weeks either in the 4-week period preceding or succeeding 3 months (ie, sustained over the period minimum 2 months to end of 3 months, or end of 3 months to end of 4 months).

CONTACTS AND LOCATIONS:
Locations (1):
- Institute of Hematology & Blood Diseases Hospital, Chinese Academy of Medical Sciences & Peking Union Medical College, Tianjin, Tianjin Municipality, China

IPD SHARING:
Plan to Share IPD: Undecided